CLINICAL TRIAL: NCT05779891
Title: Comparative Effects of Mulligan Straight Leg Raise Technique Versus Slump Stretching on Pain, Disability and Hip Range of Motion in Patients With Chronic Low Back Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahreen Anwar (Other)
Responsible Party: Sponsor-Investigator, Sahreen Anwar, Dr, Riphah International University
Organization: Riphah International University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC_FSD_00324
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group A (Experimental)
  Interventions: Other: Mulligan Traction Straight Leg Raise Technique
- Interventional Group B (Active Comparator)
  Interventions: Other: Slump Stretching

INTERVENTIONS:
Other: Mulligan Traction Straight Leg Raise Technique — The individuals in the Group A will be receive hot pack at lower back for 10 minutes followed by ultrasound at 1.5w/cm2 for 10 minutes. The treatment will be preceded by Mulligan straight leg raise technique . Three repetitions of Mulligan's Traction Straight Leg Raise will be done with 7 seconds hold and 5 seconds relax time. The total treatment protocol will be 30 minutes.
  Arms: Interventional Group A
Other: Slump Stretching — The individuals in the Group B will be receive hot pack at lower back for 10 minutes followed by ultrasound at 1.5w/cm2 for 10 minutes. The treatment will be preceded by Slump Stretching technique. Five repetitions of Slump stretching technique will be done with 30 seconds hold and 5 seconds relax time. The total treatment protocol will be 30 minutes
  Arms: Interventional Group B

SUMMARY:
The goal of this clinical trial is to examine the effect of mulligan straight leg raise versus slump stretching on pain, disability and hip range of motion in patient with low back pain. . Convenient sampling technique will be used to enroll the patients. Patients will be inquire into basis of pre formulated eligibility criteria. Written Consent will be taken from each patient before starting interventional sessions. Sample size of this study will consist on the participants who will qualify for both inclusion an exclusion criteria. Both groups will receive ultrasonic therapy and hot pack therapy as baseline treatment. Group A will receive mulligan straight leg raise and group B will receive slump stretching. The assessment of patients will be done at baseline, 4th and 8th week. The outcomes from patients will be calculated by using Visual Analogue Scale (VAS), Goniometer and ODI. The comparison between pre-treatment and post-treatment data will be done after 8th week. Data will be analyzed through SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have active positive knee extension test(APKET).
* Patient having low back pain for more than 3 months.
* Patients who have been sitting for three hours.

Exclusion Criteria:

* Any active infection, tumor, tuberculosis.
* History of trauma.
* Subject with intervertebral disc prolapse.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-06-07 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Low Back Pain | 8 weeks
  Pain will be assessed by using Numerical Pain Rating Scale
Range of motion at hip joint | 8 weeks
  Range of motion will be assessed by using Goniometer
Disability related to back pain | 8 weeks
  Disability will be assessed by using Owestry Disability Index

CONTACTS AND LOCATIONS:
Locations (1):
- District Headquarters Hospital, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No